CLINICAL TRIAL: NCT06203093
Title: Charcot-Marie-Tooth Disease (CMT) Biological Sample Collection for IPSC Generation and Biobanking
Status: Recruiting | Type: Observational
Sponsor: New York Stem Cell Foundation Research Institute (Other)
Collaborators: Charcot-Marie-Tooth Association (Other)
Responsible Party: Sponsor
Other Study IDs: 10-009
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-07

CONDITIONS: Charcot-Marie-Tooth Disease; Healthy
Keywords: Charcot-Marie-Tooth
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsy (2-3mm) and/or blood (up to 50 mL); saliva; excess/leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Charcot-Marie-Tooth Disease: Subjects in this group will have a diagnosis of Charcot-Marie-Tooth Disease.
  Interventions: Other: Biological Sample Collection
- Healthy Control: Subjects in this group will serve as healthy controls.
  Interventions: Other: Biological Sample Collection

INTERVENTIONS:
Other: Biological Sample Collection — Skin biopsy (2-3mm) and/or blood (up to 50mL); saliva; excess/leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure).

SUMMARY:
The New York Stem Cell Foundation (NYSCF) Research Institute is performing this research to accelerate Charcot-Marie-Tooth disease research and drug development by using cells from the body (such as skin or blood cells) to make stem cells and other types of cells, conduct research on the samples, perform genetic testing, and/or store the samples for future use.

Through this research, researchers hope to identify future treatments or even cures for Charcot-Marie-Tooth disease.

DETAILED DESCRIPTION:
Researchers at the New York Stem Cell Foundation (NYSCF) Research Institute study diverse diseases, conditions, and traits by creating stem cells from biological samples. These "pluripotent" stem cells can become any cell in the human body, including cells that may be difficult, invasive, or impossible to obtain directly.

Additionally, researchers perform genetic testing to learn more about DNA, a material in most cells that contains instructions for the body's development and functions (such as traits like eye color and risk of certain diseases). A piece of DNA that determines the specific role of a cell is called a "gene." If the instructions in a gene are abnormal, this can lead to disease.

Participation in the study involves: (1) completion of health questionnaires, (2) providing a skin and/or blood sample from which stem cells may be created, (3) collection of a saliva sample for genetic analysis, and (4) possible future followup to provide additional information or learn about other research studies.

This study is not a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 years or older.
* Diagnosis of Charcot-Marie-Tooth (CMT) disease or healthy controls.
* Adults must provide written informed consent unless physical limitations preclude signing.
* Minors undergoing skin collection for research purposes must have a CMT diagnosis and must participate with parent/guardian consent.
* Minors undergoing blood and/or saliva collection for research purposes or who transfer biological samples from a procedure outside the research may have a CMT diagnosis or serve as a healthy control and may participate with parent/guardian consent.

Exclusion Criteria:

* Wards of the state.
* For prospective skin samples: history of keloid formation, coagulation disorder, allergy to the anesthetic, or anticoagulation use that precludes sample collection.
* For prospective blood samples: coagulation disorder or other medical conditions that increase the risks associated with blood collection.
* For all prospective sample collections: Subjects who refuse to adhere to NYSCF's and/or a collaborating site's safety protocols will be excluded. Subjects with an AIDS diagnosis and CD4 count of less than 200 cells per microliter of blood will be excluded due to increased risk of infection.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a Charcot-Marie-Tooth (CMT) diagnosis. Individuals without a condition to serve as healthy controls (a comparison group for CMT subjects).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Biobank | Baseline
  Establishment of a bank of stem cell lines and associated information to advance understanding of the biology, etiology, manifestations, progression, risk factors, genetic underpinnings, and treatment of Charcot-Marie-Tooth diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Andres-Martin, Principal Investigator — New York Stem Cell Foundation Research Institute
Locations (1):
- New York Stem Cell Foundation Research Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No